CLINICAL TRIAL: NCT03984110
Title: The Use of a Combination of Ozurdex and Eylea Versus Eylea Monotherapy for Diabetic Macular Edema: A Prospective, Comparative Trial
Brief Title: One Year Trial Evaluating Safety of Ozurdex With Eylea
Acronym: COED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Retina Associates (Other)
Collaborators: The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRA-COED-19-001
Record Dates: First submitted 2019-06-11; First posted 2019-06-12 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Calcium Dobesilate; Dexamethasone; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combination of Ozurdex and Eylea (Experimental): Eyes receiving intravitreal injection of Ozurdex every 3 months (as needed per protocol) and intravitreal injection of Eylea every month (as needed per protocol)
  Interventions: Drug: Ozurdex; Drug: Eylea
- Eylea Monotherapy (Active Comparator): Eyes receiving intravitreal injection of Eylea every month (as needed per protocol)
  Interventions: Drug: Eylea

INTERVENTIONS:
Drug: Ozurdex — Intravitreal injection
  Other Names: dexamethasone implant
  Arms: Combination of Ozurdex and Eylea
Drug: Eylea — Intravitreal injection
  Other Names: aflibercept

SUMMARY:
One Year Trial Evaluating Safety of Ozurdex With Eylea (COED)

DETAILED DESCRIPTION:
In this study, the investigators aim to compare the effects of combined use of intravitreal injections of Ozurdex every three3 months and monthly Eylea/aflibercept to monthly intravitreal injections of aflibercept alone as measured by improvement in central subfield thickness from baseline at Week 48 in eyes with center-involving Diabetic Macular Edema and best-corrected visual acuity of 20/40 or worse

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or 2 diabetic patients
2. At least 18 years of age, understands the language of the informed consent, and is willing and able to provide written informed consent before any study procedures
3. Pseudophakic or phakic lens status with intact posterior lens capsule and/or Nd: Yttrium Aluminum Garnet (YAG) laser capsulotomy that in the investigator's opinion is not likely to permit dislocation of Ozurdex implant into the anterior chamber
4. Center-involving DME > 300 µm
5. Baseline BCVA between 20/40 - 20/320
6. Eyes with intraocular pressure (IOP) ≤ 21 and / or treatment with < 2 topical IOP-lowering medications (eyes with history of previous angle -closure or similar conditions that have been successfully treated with either laser or surgical intervention are allowed as long as the visual fields and optic nerves have been stable for > 1 year prior to study entry and the patient has been and can be safely dilated)

Exclusion Criteria:

1. Patients with active or suspected ocular or periocular infections including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
2. Patients with known hypersensitivity to any components of Eylea or Ozurdex
3. Patient has suffered from a stroke or transient ischemic attack (TIA) in the last 6 months
4. Patients using topical anti-inflammatory medication for the duration of the study
5. Patients with Anterior Chamber Intraocular Lens (ACIOL) and rupture of the posterior lens capsule
6. Prior panretinal photocoagulation or macular laser treatments within 90 days of screening
7. Previous vitrectomy
8. Any ocular condition that in the opinion of the investigator would not permit improvement of visual acuity with resolution of DME (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates and/or poor foveal architecture suggestive of photoreceptor loss)
9. Patients with retinal diseases other than diabetes that can affect macular edema
10. Eyes with a history of advanced glaucoma (optic nerve head change consistent with glaucoma damage and/or glaucomatous visual field loss), uncontrolled ocular hypertension (baseline IOP > 21 mmHg despite use of ≥ 2 topical IOP-lowering medication)
11. Eyes with a history of steroid response (i.e., increase of ≥ 5 mmHg IOP following topical steroid treatment)
12. Female patients who are pregnant or breastfeeding
13. Patients who are unable to attend scheduled follow-up visits throughout the 24-week study
14. Any intravitreal anti-Vascular Endothelial Growth Factor (VEGF) treatment to study eye within 3 months prior to Day 1
15. Use of systemic steroid, anti-VEGF or pro-VEGF treatment within 4 months prior to enrollment or anticipated use during the study (these drugs are prohibited from use during the study)
16. History of any previous treatment in the study eye with an ocular corticosteroid implant (eg Iluvien, Ozurdex, Retisert)
17. Has scarring from laser photocoagulation in the study eye that would compromise Visual Acuity (VA); or scarring or abnormality from other macular condition, in the investigator's medical judgement, would limit VA (such as an epiretinal membrane or macular hole)
18. Has significant media opacity precluding evaluation of retina and vitreous in the study eye. This includes cataract that is felt to be a major contributor to reduced visual acuity and/or likely to undergo surgical repair within 3 months of randomization.
19. Has any uncontrolled systemic disease that, in the opinion of the Investigator, would preclude participation in the study (eg, infection, uncontrolled elevated blood pressure, cardiovascular disease, poor glycemic control) or put the subject at risk due to study treatment or procedures
20. Has had a myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 1 month before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Central Subfield Thickness (CST) | 48 weeks
  Change in Central Subfield Thickness (CST) on Spectral Domain-Optical Coherence Tomography (SD-OCT)

SECONDARY OUTCOMES:
CST | 12 weeks, 24 weeks, and 36 weeks
  Change in CST
Best Corrected Visual Acuity (BCVA) | 12 weeks, 24 weeks, 36 weeks, and 48 weeks
  Change in Best Corrected Visual Acuity (BCVA)
Number of additional Intravitreal Therapy (IVT) aflibercept injections required over 48 weeks | 48 weeks
  Number of additional Intravitreal Therapy (IVT) aflibercept injections required over 48 weeks
Monthly mean changes from baseline in BCVA | 48 weeks
  Monthly mean changes from baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study (ETDRS) letters read
Monthly mean changes from baseline in CST | 48 weeks
  Monthly mean changes from baseline in CST as measured by SD-OCT

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan M Abbey, MD, Principal Investigator — Texas Retina Associates
Locations (1):
- Texas Retina Associates, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No